CLINICAL TRIAL: NCT02085408
Title: Phase III Randomized Trial of Clofarabine as Induction and Post-Remission Therapy vs. Standard Daunorubicin &Amp; Cytarabine Induction and Intermediate Dose Cytarabine Post-Remission Therapy, Followed by Decitabine Maintenance vs. Observation in Newly-Diagnosed Acute Myeloid Leukemia in Older Adults (Age >/= 60 Years)
Brief Title: Clofarabine or Daunorubicin Hydrochloride and Cytarabine Followed By Decitabine or Observation in Treating Older Patients With Newly Diagnosed Acute Myeloid Leukemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ECOG-ACRIN Cancer Research Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: Eastern Cooperative Oncology Group (Network)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E2906; NCI-2011-01992 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000659585; E2906 (Other: Eastern Cooperative Oncology Group); E2906 (Other: CTEP); U10CA021115 (NIH); NCT01041703 (obsolete NCT alias)
Record Dates: First submitted 2014-03-11; First posted 2014-03-12 (Estimated); Results first posted 2023-03-09 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-11

CONDITIONS: Acute Myeloid Leukemia With Multilineage Dysplasia Following Myelodysplastic Syndrome; Adult Acute Megakaryoblastic Leukemia (M7); Adult Acute Minimally Differentiated Myeloid Leukemia (M0); Adult Acute Monoblastic Leukemia (M5a); Adult Acute Monocytic Leukemia (M5b); Adult Acute Myeloblastic Leukemia With Maturation (M2); Adult Acute Myeloblastic Leukemia Without Maturation (M1); Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Del(5q); Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); Adult Acute Myelomonocytic Leukemia (M4); Adult Erythroleukemia (M6a); Adult Pure Erythroid Leukemia (M6b); Secondary Acute Myeloid Leukemia; Untreated Adult Acute Myeloid Leukemia
Keywords: acute myeloid leukemia; Clofarabine; Daunorubicin; Cytarabine; Decitabine
MeSH Terms: conditions — Leukemia, Megakaryoblastic, Acute; Leukemia, Monocytic, Acute; Leukemia, Myeloid, Acute; Congenital Abnormalities; Leukemia, Myelomonocytic, Acute; Leukemia, Erythroblastic, Acute | interventions — Daunorubicin; Cytarabine; Clofarabine; Decitabine; Observation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- A (Induction:daunorubicin/cytarabine; consolidation:cytarabine; maintenance:observation/transplant) (Active Comparator): See Detailed Description
  Interventions: Drug: Daunorubicin; Drug: Cytarabine; Other: Observation; Procedure: Allogeneic hematopoietic stem cell transplantation
- B (Induction: clofarabine; Consolidation: clofarabine; Maintenance: decitabine or transplant) (Experimental): See Detailed Description
  Interventions: Drug: Clofarabine; Drug: Decitabine; Procedure: Allogeneic hematopoietic stem cell transplantation

INTERVENTIONS:
Drug: Daunorubicin — Given IV
  Other Names: Daunomycin; Cerubidine; Rubidomycin
  Arms: A (Induction:daunorubicin/cytarabine; consolidation:cytarabine; maintenance:observation/transplant)
Drug: Cytarabine — Given IV
  Other Names: Ara-C; Arabinosyl; Cytosar-U; cytosine arabinoside
  Arms: A (Induction:daunorubicin/cytarabine; consolidation:cytarabine; maintenance:observation/transplant)
Drug: Clofarabine — Given IV
  Other Names: CLOLAR; Cl-F-Ara-A, 2-chloro-9-(2-deoxy-2-fluoro-β-Darabinofuranosyl)adenine
  Arms: B (Induction: clofarabine; Consolidation: clofarabine; Maintenance: decitabine or transplant)
Drug: Decitabine — Given IV
  Other Names: Dacogen®; 5-aza-2'-deoxycytidine; 5-aza-CdR
  Arms: B (Induction: clofarabine; Consolidation: clofarabine; Maintenance: decitabine or transplant)
Other: Observation — Undergo clinical observation
  Arms: A (Induction:daunorubicin/cytarabine; consolidation:cytarabine; maintenance:observation/transplant)
Procedure: Allogeneic hematopoietic stem cell transplantation — Patients with an HLA-identical donor proceed to allogeneic stem cell transplantation.
  Other Names: AlloSCT

SUMMARY:
This randomized phase III trial studies clofarabine to see how well it works compared with daunorubicin hydrochloride and cytarabine when followed by decitabine or observation in treating older patients with newly diagnosed acute myeloid leukemia. Drugs used in chemotherapy, such as clofarabine, daunorubicin hydrochloride, cytarabine, and decitabine, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more cancer cells. It is not yet known which chemotherapy regimen is more effective in treating acute myeloid leukemia.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the effect of clofarabine induction and consolidation therapy on overall survival in comparison with standard therapy (daunorubicin [daunorubicin hydrochloride] & cytarabine) in newly-diagnosed acute myeloid leukemia (AML) patients age >= 60 years.

SECONDARY OBJECTIVES:

I. To evaluate complete remission (CR) rates, duration of remission, and toxicity/treatment-related mortality of clofarabine in comparison with standard therapy (daunorubicin & cytarabine) in newly-diagnosed AML patients age >= 60 years.

II. To evaluate the feasibility of consolidation with reduced-intensity conditioning and allogeneic hematopoietic stem cell transplantation from human leukocyte antigen (HLA)-identical donors in patients who achieve a response to induction therapy, including the incidence of successful engraftment, acute and chronic graft-versus-host disease, transplant-related mortality, and its impact on overall survival in comparison to patients receiving chemotherapy.

III. To evaluate the duration of remission and disease-free survival of patients in complete remission following completion of consolidation therapy who are subsequently randomized to receive scheduled low-dose decitabine maintenance in comparison with observation.

IV. To perform expression and methylation profiling on all patients receiving decitabine and to correlate their integrated epigenetic signatures with response to decitabine.

V. To examine the epigenetic profiles of remission marrow in patients randomized to observation vs. decitabine to determine whether epigenetic signature of apparently morphologically normal bone marrow is predictive of relapse or response to decitabine maintenance.

VI. To explore the possible association of response to clofarabine with ABC-transporter P-glycoprotein (Pgp).

VII. To assess the intensity of expression of CXC chemokine receptor type 4 (CXCR4) on diagnostic leukemia cells and to correlate this parameter with other established prognostic factors.

VIII. To assess the entire spectrum of somatic mutations and affected pathways at diagnosis of AML and elucidate the association between gene mutation and outcome.

IX. To examine the impact of smoking, obesity, regular acetaminophen use, regular aspirin use, benzene exposure, living in a rural/farm environment and some other underlying exposures and lifestyle factors associated with AML development on overall survival (OS).

X. To investigate potential correlative results between array comparative genomic hybridization (CGH) findings and acute myeloid leukemia patient characteristics.

TERTIARY OBJECTIVES:

I. To compare health-related quality of life (QOL) (physical, functional, leukemia-specific well-being) and fatigue in elderly AML patients receiving standard induction therapy with those receiving clofarabine.

II. To measure the change in health-related QOL that occurs over time (within treatment groups).

III. To comprehensively assess patient function at the time of study enrollment.

IV. To determine if components of a comprehensive geriatric assessment or QOL scales predict ability to complete AML treatment.

V. To describe the impact of transplant on QOL in AML patients above age 60.

OUTLINE:

INDUCTION THERAPY: Patients are randomized to 1 of 2 treatment arms.

ARM A (STANDARD THERAPY): Patients receive daunorubicin hydrochloride at 60 mg/m^2 intravenously (IV) over 10-15 minutes on days 1-3 and cytarabine at 100 mg/m^2 IV continuously on days 1-7. Patients with residual disease or those who do not achieve an aplastic bone marrow on day 12-14 (i.e., < 5% blasts and < 20% cellularity or markedly/moderately hypocellular) may receive a second course of induction therapy beginning no sooner than day 14.

ARM B: Patients receive clofarabine at 30 mg/m^2 IV over 1 hour on days 1-5. Patients with residual disease or those who do not achieve an aplastic bone marrow on day 12-14 (i.e., < 5% blasts and < 20% cellularity or markedly/moderately hypocellular) may receive a second course of induction therapy beginning no sooner than day 21 and no later than day 56.

Patients who achieve a complete remission (CR) or CR with incomplete marrow recovery (CRi) after induction therapy proceed to consolidation therapy (Arms C and D). Patients who are 60-69 years of age who achieve a "morphologic leukemia-free state" after induction therapy and who have an HLA-identical donor proceed to allogeneic stem cell transplantation.

CONSOLIDATION THERAPY: Beginning within 60 days after documentation of CR or CRi, patients receive consolidation therapy in the same arm they were randomized to for induction therapy.

ARM C (STANDARD THERAPY): Patients receive cytarabine at 1500 mg/m^2 IV over 1 hour once or twice daily on days 1-6. Treatment repeats every 4-6 weeks for 2 courses.

ARM D: Patients receive clofarabine at 20 mg/m^2 IV over 1 hour on days 1-5. Treatment repeats every 4-6 weeks for 2 courses.

Patients who remain in CR after completion of consolidation therapy are randomized to one of the two maintenance therapy arms (Arms E and F).

MAINTENANCE THERAPY: Beginning within 60 days after completion of consolidation therapy, patients receive maintenance therapy and are randomized to 1 of 2 arms. Patients not eligible for randomization to decitabine maintenance after recovery from consolidation will be followed according to Arm E.

ARM E: Patients undergo observation monthly for 12 months.

ARM F: Patients receive decitabine at 20 mg/m^2 IV over 1 hour on days 1-3. Treatment repeats every 4 weeks for 12 months the absence of unacceptable toxicity.

ALLOGENEIC STEM CELL TRANSPLANTATION WITH REDUCED-INTENSITY CONDITIONING REGIMEN (Arm G): Patients begin reduced-intensity conditioning 30-90 days after the initiation of induction therapy.

CONDITIONING REGIMEN: Patients receive fludarabine phosphate at 30 mg/m^2 IV over 30 minutes on days -7 to -3, busulfan at 0.8 mg/kg IV over 2 hours every 6 hours on days -4 and -3 (for a total of 8 doses), and anti-thymocyte globulin at 2.5 mg/kg/day IV over 4-6 hours on days -4 to -2.

TRANSPLANTATION: Patients undergo allogeneic peripheral blood stem cell transplantation on day 0.

After completion of study treatment, patients are followed up every 3 months for 4 years, every 6 months for 1 year, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria for Step 1 (Induction):

* Sexually active males must be strongly advised to use an accepted and effective method of contraception
* Aspartate aminotransferase (AST), alanine aminotransferase (ALT), total bilirubin =< grade 1
* Newly-diagnosed AML patients according to World Health Organization (WHO) classification who are considered candidates for intensive chemotherapy based upon examination of peripheral blood or bone marrow aspirate specimens or touch preparations of the bone marrow biopsy obtained within two weeks prior to randomization; a bone marrow aspirate is required for enrollment; however, on occasion there is discordance between percentage of myeloblasts on the differential of the peripheral blood or aspirate; the peripheral blood criteria are sufficient for diagnosis; confirmatory immunophenotyping will be performed centrally
* ECOG performance status (PS) 0-3 (restricted to ECOG PS 0-2 if >= 70 years of age)
* Patients with secondary AML are eligible for enrollment onto the trial; secondary AML is defined as AML that has developed in a person with a history of antecedent blood count abnormalities, or myelodysplastic syndrome (MDS), or a myeloproliferative disorder (excluding chronic myeloid leukemia); or a history of prior chemotherapy or radiation therapy for a disease other than AML
* Total serum bilirubin =< 1.5 times upper limit of normal (ULN) (=< grade 1); if total bilirubin is 2 to 3 mg/dL, but direct bilirubin is normal, then the patient will be considered eligible
* Patients with a serum creatinine > 1 are eligible if they have a calculated glomerular filtration rate (GFR) of >= 60 ml/min (i.e. class I or class II chronic kidney disease ) using the Modification of Diet in Renal Disease (MDRD) formula

  * Note: Daily creatinine and MDRD formula are only for the 1st induction cycle
* Cardiac ejection fraction >= 45% or within institutional normal limits; a nuclear medicine gated blood pool examination is preferred; a two-dimensional (2-D) echocardiogram (ECHO) scan is acceptable if a calculated ejection fraction is obtained and follow-up measurement of the cardiac ejection fraction will also be performed by echocardiography; measurement of cardiac ejection fraction should be within two weeks prior to receiving treatment

  * NOTE: when a multi gated acquisition scan (MUGA) or echocardiogram cannot be obtained due to weekend or holiday, then patients may be enrolled provided there is no history of significant cardiovascular disease and a measurement of cardiac ejection fraction will be performed within 5 days of study enrollment
* Patients with suspected central nervous system (CNS) involvement should undergo lumbar puncture
* Cytogenetic analysis must be performed from diagnostic bone marrow (preferred) or if adequate number of circulating blasts (>10^9/l) from peripheral blood
* HLA typing should be performed at registration, if possible
* Diagnostic bone marrow and peripheral blood specimens must be submitted for immunophenotyping and selected molecular testing

Exclusion Criteria for Step 1 (Induction):

* Concurrent active malignancy for which they are receiving treatment (other than myelodysplastic syndromes [MDS])
* Active, uncontrolled infection
* Acute promyelocytic leukemia (APL) confirmed either by the presence of t(15;17)(q22;q21) or promyelocytic leukemia (PML)/retinoic acid receptor (RAR) alpha transcripts
* Blastic transformation of chronic myelogenous leukemia
* Prior therapy of MDS with decitabine, low-dose cytarabine, or azacitidine
* Prior chemotherapy for AML with the exception of hydroxyurea for increased blast count or leukapheresis for leukocytosis
* Documented CNS involvement
* Previous treatment for antecedent hematological disorders (AHD) with 5-azacitidine, decitabine, or low dose cytarabine
* Human immunodeficiency virus (HIV) infection

Inclusion Criteria for Step 2 (Consolidation)

* NOTE: All patients achieving complete remission (CR) or complete remission with incomplete blood count recovery (CRi) will receive consolidation when fit
* NOTE: Patients proceeding to transplant are allowed up to one cycle of consolidation treatment
* Consolidation cycle 1 must commence within sixty days of the bone marrow aspirate and biopsy that confirmed the presence of a CR or CRi
* Patients must have achieved a CR or CRi (or morphologic leukemia-free state for those patients proceeding to Arm G transplant)
* Patients who have achieved a CR or CRi must have maintained peripheral blood evidence of a CR or CRi
* ECOG performance status of 0-2
* Patients must have resolved any serious infectious complications related to induction

  * NOTE: Patients with an HLA-matched donor and proceeding to transplant will be allowed up to one cycle of consolidation treatment
* Any significant medical complications related to induction must have resolved
* Patients must have a creatinine and AST =< grade 1 within 48 hours prior to registration

Inclusion Criteria for Step 3 (Maintenance):

* Maintenance should commence within 60 days of recovery of peripheral blood counts after consolidation cycle 2; patients must begin consolidation cycle 2 within 60 days of recovery to be eligible for further therapy
* Patients must have maintained peripheral blood evidence of a remission and must have a CR or CRi, confirmed on restaging bone marrow (BM) aspirate and biopsy and cytogenetic analysis
* ECOG performance status of 0 -2
* Patients must have resolved any serious infectious complications related to consolidation cycle 2
* Any significant medical complications related to consolidation cycle 2 must have resolved
* Total serum bilirubin =< 1.5 x ULN

  * NOTE: if total bilirubin is 2-3 mg/dL, but direct bilirubin is normal, then the patient will be considered eligible
* Serum creatinine =< grade 1
* The absolute neutrophil count (ANC) must be > 1000 mm^3 prior to starting every cycle of treatment with decitabine; decitabine may be delayed for up to 4 weeks between cycles (i.e. may be administered as infrequently as every (q) 8 weeks) while waiting for counts to recover
* The platelet count must be > 75,000 mm^3 prior to starting every cycle of treatment with decitabine; decitabine may be delayed for up to 4 weeks between cycles (i.e. may be administered as infrequently as every (q) 8 weeks) while waiting for counts to recover

Inclusion Criteria for Step 3 (Allogeneic Transplantation):

* Patients must be > 28 days from the start of induction or re-induction chemotherapy, or from the start Consolidation Cycle 1 (if received) and < 90 days following recovery from most recent treatment; and they must have achieved and maintained a response to induction therapy (CR, CRi, or "morphologic disease-free state")
* Patients must have recovered from the effects of induction, re-induction, or consolidation chemotherapy (all toxicities =< grade I with the exception of reversible electrolyte abnormalities), and have no ongoing active infection requiring treatment
* Patients must have a total serum bilirubin =< 1.5 x ULN (grade =< 1) and a serum creatinine =< grade 1; AST <= grade 1
* An eligible HLA-identical donor (either related or unrelated) should be available; in sibling donors, low resolution HLA typing (A,B,DR) will be considered sufficient; in the case of unrelated donors, high-resolution class I and II typing (A, B, C, DRB1 and DQ) should be matched at all 10 loci; donors must be willing and able to undergo peripheral blood progenitor mobilization

  * HLA-identical sibling (6/6): the donor must be determined to be an HLA-identical sibling (6/6) by serologic typing for class (A, B) and low resolution molecular typing for class II (DRB1)
  * Matched unrelated donor (10/10): high resolution molecular typing at the following loci is required: HLA-A, -B, -C, -DRBL, and -DQB1
  * NOTE: for matched donors - will allow select 1 antigen mismatched sibling donors and unrelated donors in accordance with site institutional standard, as long as matched at HLA-A, HLA-B, HLA-C, and DRB1, and with advanced discussion/approval by the Study Chair and the bone marrow transplant (BMT) co-chair
* Patients must be considered reliable enough to comply with the medication regimen and follow-up, and have social support necessary to allow this compliance
* Patients must have a cardiac ejection fraction of >= 40%, or within institutional normal limits; a nuclear medicine gated blood pool examination is preferred; a 2-D ECHO scan is acceptable if a calculated ejection fraction is obtained and follow-up measurement of the cardiac ejection fraction will also be performed by echocardiography; measurement of cardiac ejection fraction should be within two weeks prior to allogeneic transplantation
* Diffusion capacity of carbon monoxide (DLCO) > 40% with no symptomatic pulmonary disease

Exclusion Criteria for Step 3 (Allogeneic Transplantation):

* Hypersensitivity to Escherichia (E.) coli-derived products
* Human immunodeficiency virus (HIV) infection; patients with immune dysfunction are at a significantly higher risk of toxicities from intensive immunosuppressive therapies

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 727 (Actual)
Dates: Start 2011-02-04 (Actual); Primary Completion 2021-02-22 (Actual); Study Completion 2022-12-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Foran, Principal Investigator — Eastern Cooperative Oncology Group
Locations (269):
- United States (266):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Arizona Cancer Center at University Medical Center North, Tucson, Arizona
  - University of Arizona Health Sciences Center, Tucson, Arizona
  - The Medical Center of Aurora, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Saint Anthony Central Hospital, Denver, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Exempla Saint Joseph Hospital, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Colorado Cancer Research Program CCOP, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Littleton Adventist Hospital, Littleton, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - Parker Adventist Hospital, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - Exempla Lutheran Medical Center, Wheat Ridge, Colorado
  - Saint Francis Hospital and Medical Center, Hartford, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - University of Florida, Gainesville, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Florida Hospital, Orlando, Florida
  - Piedmont Hospital, Atlanta, Georgia
  - Atlanta Regional CCOP, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - Saint Joseph's Hospital of Atlanta, Atlanta, Georgia
  - Georgia Regents University, Augusta, Georgia
  - Well Star Cobb Hospital, Austell, Georgia
  - John B Amos Cancer Center, Columbus, Georgia
  - Dekalb Medical Center, Decatur, Georgia
  - Piedmont Fayette Hospital, Fayetteville, Georgia
  - Gwinnett Medical Center, Lawrenceville, Georgia
  - Wellstar Kennestone Hospital, Marietta, Georgia
  - Southern Regional Medical Center, Riverdale, Georgia
  - Harbin Clinic Medical Oncology and Clinical Research, Rome, Georgia
  - Oncare Hawaii Inc-POB II, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii, Honolulu, Hawaii
  - OnCare Hawaii-Liliha, Honolulu, Hawaii
  - Kuakini Medical Center, Honolulu, Hawaii
  - Oncare Hawaii Inc-Kuakini, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Castle Medical Center, Kailua, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Kapiolani Medical Center at Pali Momi, ‘Aiea, Hawaii
  - Oncare Hawaii Inc - Kapiolani Medical Center at Pali Momi, ‘Aiea, Hawaii
  - Saint Alphonsus Regional Medical Center, Boise, Idaho
  - Saint Anthony's Health, Alton, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Saint Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital Association, Canton, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Mount Sinai Hospital Medical Center, Chicago, Illinois
  - Hematology and Oncology Associates, Chicago, Illinois
  - Northwestern University, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Eureka Hospital, Eureka, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Illinois CancerCare-Havana, Havana, Illinois
  - Mason District Hospital, Havana, Illinois
  - Hematology Oncology Associates of Illinois-Highland Park, Highland Park, Illinois
  - Hinsdale Hematology Oncology Associates Incorporated, Hinsdale, Illinois
  - Presence Saint Mary's Hospital, Kankakee, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - North Shore Hematology Oncology, Libertyville, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Mcdonough District Hospital, Macomb, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Holy Family Medical Center, Monmouth, Illinois
  - Illinois CancerCare-Monmouth, Monmouth, Illinois
  - Illinois Cancer Specialists-Niles, Niles, Illinois
  - Bromenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center Foundation, Normal, Illinois
  - Illinois CancerCare-Community Cancer Center, Normal, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Ottawa Regional Hospital and Healthcare Center, Ottawa, Illinois
  - Pekin Cancer Treatment Center, Pekin, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Proctor Hospital, Peoria, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Illinois Oncology Research Association CCOP, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Illinois Valley Hospital, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - Swedish American Hospital, Rockford, Illinois
  - Hematology Oncology Associates of Illinois - Skokie, Skokie, Illinois
  - Illinois CancerCare-Spring Valley, Spring Valley, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Saint Francis Hospital and Health Centers, Beech Grove, Indiana
  - Fort Wayne Medical Oncology and Hematology Inc - State Boulevard, Fort Wayne, Indiana
  - Franciscan St. Francis Health, Indianapolis, Indiana
  - Reid Hospital and Health Care Services, Richmond, Indiana
  - McFarland Clinic, Ames, Iowa
  - Siouxland Hematology Oncology Associates, Sioux City, Iowa
  - Mercy Medical Center-Sioux City, Sioux City, Iowa
  - Saint Luke's Regional Medical Center, Sioux City, Iowa
  - University of Kentucky, Lexington, Kentucky
  - Norton Health Care Pavilion - Downtown, Louisville, Kentucky
  - Ochsner Clinic Foundation-Baton Rouge, Baton Rouge, Louisiana
  - Ochsner Baptist Medical Center, New Orleans, Louisiana
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Harold Alfond Center for Cancer Care, Augusta, Maine
  - Eastern Maine Medical Center, Bangor, Maine
  - Johns Hopkins University, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Union Hospital of Cecil County, Elkton, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Caritas Saint Elizabeth's Medical Center, Brighton, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Michigan Cancer Research Consortium Community Clinical Oncology Program, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - Mecosta County Medical Center, Big Rapids, Michigan
  - Oakwood Hospital, Dearborn, Michigan
  - Wayne State University, Detroit, Michigan
  - Saint John Hospital and Medical Center, Detroit, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Genesys Regional Medical Center-West Flint Campus, Flint, Michigan
  - Genesys Regional Medical Center, Grand Blanc, Michigan
  - Grand Rapids Clinical Oncology Program, Grand Rapids, Michigan
  - Saint Mary's Health Care, Grand Rapids, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - Allegiance Health, Jackson, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - Mercy Health Partners-Mercy Campus, Muskegon, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Saint Joseph Mercy Port Huron, Port Huron, Michigan
  - Spectrum Health Reed City Hospital, Reed City, Michigan
  - Saint Mary's of Michigan, Saginaw, Michigan
  - Providence Hospital, Southfield, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Sanford Clinic North-Bemidgi, Bemidji, Minnesota
  - Essentia Health Saint Joseph's Medical Center, Brainerd, Minnesota
  - Essentia Health Duluth Clinic CCOP, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Lake Region Healthcare Corporation-Cancer Care, Fergus Falls, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Saint Louis Cancer and Breast Institute-South City, St Louis, Missouri
  - Saint Louis University Hospital, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Saint John's Mercy Medical Center, St Louis, Missouri
  - Saint Louis-Cape Girardeau CCOP, St Louis, Missouri
  - Montana Cancer Consortium CCOP, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies PC, Billings, Montana
  - Billings Clinic, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Northern Montana Hospital, Havre, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Glacier Oncology PLLC, Kalispell, Montana
  - Kalispell Medical Oncology, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Montana Cancer Specialists, Missoula, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Nevada Cancer Research Foundation CCOP, Las Vegas, Nevada
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Winthrop University Hospital, Mineola, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Rochester, Rochester, New York
  - Park Ridge Hospital Breast Health Center, Hendersonville, North Carolina
  - Kinston Medical Specialists PA, Kinston, North Carolina
  - Roger Maris Cancer Center, Fargo, North Dakota
  - Sanford Clinic North-Fargo, Fargo, North Dakota
  - Sanford Medical Center-Fargo, Fargo, North Dakota
  - Summa Akron City Hospital, Akron, Ohio
  - Akron General Medical Center, Akron, Ohio
  - Summa Barberton Hospital, Barberton, Ohio
  - Aultman Health Foundation, Canton, Ohio
  - The Jewish Hospital, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Health Center, Dayton, Ohio
  - Dayton CCOP, Dayton, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Saint Rita's Medical Center, Lima, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Clinton Memorial Hospital, Wilmington, Ohio
  - Greene Memorial Hospital, Xenia, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Columbia River Oncology Program, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Lehigh Valley Hospital, Allentown, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazelton, Hazleton, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - Abramson Cancer Center of The University of Pennsylvania, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - Mount Nittany Medical Center, State College, Pennsylvania
  - Geisinger Wyoming Valley, Wilkes-Barre, Pennsylvania
  - York Hospital, York, Pennsylvania
  - AnMed Health Cancer Center, Anderson, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Carolina Blood and Cancer Care Associates PA-Lancaster, Lancaster, South Carolina
  - Carolina Blood and Cancer Care Associates PA, Rock Hill, South Carolina
  - Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Upstate Carolina CCOP, Spartanburg, South Carolina
  - Sanford Cancer Center-Oncology Clinic, Sioux Falls, South Dakota
  - Medical X-Ray Center, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Erlanger Medical Center, Chattanooga, Tennessee
  - Jackson-Madison County General Hospital, Jackson, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Northwest Cancer Specialists, Vancouver, Washington
  - West Virginia University Charleston, Charleston, West Virginia
  - West Virginia University, Morgantown, West Virginia
  - Green Bay Oncology at Saint Vincent Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital, Green Bay, Wisconsin
  - Green Bay Oncology Limited at Saint Mary's Hospital, Green Bay, Wisconsin
  - Saint Mary's Hospital, Green Bay, Wisconsin
  - Gundersen Lutheran, La Crosse, Wisconsin
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Holy Family Memorial Hospital, Manitowoc, Wisconsin
  - Bay Area Medical Center, Marinette, Wisconsin
  - Froedtert and the Medical College of Wisconsin, Milwaukee, Wisconsin
  - D N Greenwald Center, Mukwonago, Wisconsin
  - Oconomowoc Memorial Hospital-ProHealth Care Inc, Oconomowoc, Wisconsin
  - Saint Nicholas Hospital, Sheboygan, Wisconsin
  - Waukesha Memorial Hospital - ProHealth Care, Waukesha, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Rocky Mountain Oncology, Casper, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming
- Mayo Clinic Methodist Hospital, Nagpur, India
- Israel (2):
  - Rambam Medical Center, Haifa
  - Shaare Zedek Medical Center, Jerusalem

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data may be made available upon request as per the ECOG-ACRIN Data Sharing Policy.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was activated on December 28, 2010, accrued its first patient on February 4, 2011, and closed on January 24, 2019 for a total of 727 patients enrolled.
Groups:
- A (Step 1:Daunorubicin/Cytarabine; Step 2:Cytarabine; Step 3: Observation/Decitabine/Transplant): Patients in Arm A who achieve a CR or CRi after induction therapy (Step 1) proceed to consolidation therapy (Step 2 - Cytarabine; Arm C).
  Patients who remain in CR or CRi after completion of consolidation therapy are randomized to one of the two maintenance therapy (Step 3) arms (Arm E: observation or Arm F: Decitabine).
  Patients who achieve a "morphologic leukemia-free state" after induction therapy in Arm A and who have an HLA-identical donor proceed to consolidation therapy (Cytarabine; Arm C) followed by allogeneic stem cell transplantation (Arm G).
- B (Step 1: Clofarabine; Step 2: Clofarabine; Step 3: Observation/Decitabine/Transplant): Patients in Arm B who achieve a CR or CRi after induction therapy (Step 1) proceed to consolidation therapy (Step 2 - Clofarabine; Arm D).
  Patients who remain in CR or CRi after completion of consolidation therapy are randomized to one of the two maintenance therapy (Step 3) arms (Arm E: observation or Arm F: Decitabine).
  Patients who achieve a "morphologic leukemia-free state" after induction therapy in Arm B and who have an HLA-identical donor proceed to consolidation therapy (Clofarabine; Arm D) followed by allogeneic stem cell transplantation (Arm G).
Period: Step 1: Induction
Arm/Group | A (Step 1:Daunorubicin/Cytarabine; Step 2:Cytarabine; Step 3: Observation/Decitabine/Transplant) | B (Step 1: Clofarabine; Step 2: Clofarabine; Step 3: Observation/Decitabine/Transplant)
Started | 363 | 364
Adverse Event Data Available | 356 | 360
Donor Information Available | 191 | 195
Completed | 227 | 225
Not Completed | 136 | 139
Not completed — Disease Progression | 19 | 19
Not completed — Adverse Event | 18 | 17
Not completed — Death | 33 | 30
Not completed — Withdrawal by Subject | 16 | 8
Not completed — Alternative Therapy | 15 | 19
Not completed — Complicating Disease | 2 | 3
Not completed — Other | 27 | 39
Not completed — Never started treatment | 6 | 4
Period: Step 2: Consolidation
Arm/Group | A (Step 1:Daunorubicin/Cytarabine; Step 2:Cytarabine; Step 3: Observation/Decitabine/Transplant) | B (Step 1: Clofarabine; Step 2: Clofarabine; Step 3: Observation/Decitabine/Transplant)
Started | 174 | 154
Adverse Event Data Available | 170 | 148
Completed | 129 | 104
Not Completed | 45 | 50
Not completed — Disease Progression | 5 | 20
Not completed — Adverse Event | 9 | 8
Not completed — Death | 4 | 3
Not completed — Withdrawal by Subject | 8 | 5
Not completed — Alternative Therapy | 9 | 3
Not completed — Complicating Disease | 0 | 2
Not completed — Other | 6 | 6
Not completed — Never started treatment | 4 | 3
Period: Step 3: Maintenance
Arm/Group | A (Step 1:Daunorubicin/Cytarabine; Step 2:Cytarabine; Step 3: Observation/Decitabine/Transplant) | B (Step 1: Clofarabine; Step 2: Clofarabine; Step 3: Observation/Decitabine/Transplant)
Started | 103 | 89
Randomized to Observation | 35 | 26
Randomized to Decitabine | 32 | 27
Received Transplant | 36 | 36
Completed | 78 | 67
Not Completed | 25 | 22
Not completed — Disease Progression | 13 | 11
Not completed — Adverse Event | 2 | 4
Not completed — Death | 1 | 2
Not completed — Alternative Therapy | 1 | 1
Not completed — Complicating Disease | 0 | 1
Not completed — Other | 3 | 2
Not completed — Never started treatment | 5 | 1

BASELINE CHARACTERISTICS:
Population: All randomized patients are included in this analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | A (Step 1:Daunorubicin/Cytarabine; Step 2:Cytarabine; Step 3: Observation/Decitabine/Transplant) | B (Step 1: Clofarabine; Step 2: Clofarabine; Step 3: Observation/Decitabine/Transplant) | Total
Number analyzed (Participants) | 363 | 364 | 727
Age, Continuous [Median (Full Range); unit: years] | 68 [60 to 86] | 68 [60 to 85] | 68 [60 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 162 | 151 | 313
  Male | 201 | 213 | 414
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 12 | 18
  Not Hispanic or Latino | 306 | 295 | 601
  Unknown or Not Reported | 51 | 57 | 108
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 2 | 7 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 17 | 18 | 35
  White | 334 | 328 | 662
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 9 | 9 | 18

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Overall survival is defined as the time from randomization to death or date last known alive.
Time Frame: Assessed every 3 months for 4 years and then every 6 months for 1 year
Population: All randomized patients are included in this analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | A (Step 1:Daunorubicin/Cytarabine; Step 2:Cytarabine; Step 3: Observation/Decitabine/Transplant) | B (Step 1: Clofarabine; Step 2: Clofarabine; Step 3: Observation/Decitabine/Transplant)
Number analyzed (Participants) | 363 | 364
months | 12.9 [11.0 to 14.9] | 11.6 [9.8 to 14.1]
Statistical Analysis 1: Comparison: A (Step 1:Daunorubicin/Cytarabine; Step 2:Cytarabine; Step 3: Observation/Decitabine/Transplant) vs B (Step 1: Clofarabine; Step 2: Clofarabine; Step 3: Observation/Decitabine/Transplant); Test type: Superiority; Regression, Cox; Hazard Ratio (HR) = 1.1, 95% CI 2-sided [0.94 to 1.30] — Hazard ratio : clofarabine/(daunorubicin & cytarabine)

2. Secondary Outcome: Proportion of Patients With Complete Remission
Description: Patients are required to have all of the following to be considered as having a completion remission (CR).
  * Peripheral Blood Counts
    1. Neutrophil count > 1.0 x 10^9 /L
    2. Platelet count ≥ 100 x 10^9 /L
    3. Reduced hemoglobin concentration or hematocrit has no bearing on remission status
    4. Leukemic blasts must not be present in the peripheral blood
  * Bone Marrow Aspirate and Biopsy
    1. Cellularity of bone marrow biopsy must be > 20% with maturation of all cell lines
    2. < 5% blasts by morphologic review
    3. Auer rods must not be detectable
  * Extramedullary leukemia, such as CNS or soft tissue involvement, must not be present
Time Frame: Assessed every 3 months for 4 years and then every 6 months for 1 year
Population: All randomized patients are included in this analysis.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | A (Step 1:Daunorubicin/Cytarabine; Step 2:Cytarabine; Step 3: Observation/Decitabine/Transplant) | B (Step 1: Clofarabine; Step 2: Clofarabine; Step 3: Observation/Decitabine/Transplant)
Number analyzed (Participants) | 363 | 364
proportion of participants | 0.446 [0.394 to 0.499] | 0.453 [0.401 to 0.506]
Statistical Analysis 1: Comparison: A (Step 1:Daunorubicin/Cytarabine; Step 2:Cytarabine; Step 3: Observation/Decitabine/Transplant) vs B (Step 1: Clofarabine; Step 2: Clofarabine; Step 3: Observation/Decitabine/Transplant); Test type: Superiority; p = 0.94, Fisher Exact

3. Secondary Outcome: Overall Survival by Donor Status
Description: Overall survival is defined as time between achieving leukemia-free state after induction therapy to death from any cause or date last known alive. The association between overall survival and donor status was evaluated regardless of assigned treatment arms. Patients with transplant donor information (either had donor or did not have a donor) reported after achieving CR/Cri/leukemia-free state post induction therapy were included in this analysis.
Time Frame: Assessed every 3 months for 4 years and then every 6 months for 1 year
Population: Patients with transplant donor information (either had donor or did not have a donor) reported after achieving CR/Cri/leukemia-free state post induction therapy
Measure: Median (95% Confidence Interval); unit: months
Groups:
- With Transplant Donor: Patients who had transplant donor after achieving CR/Cri/leukemia-free state after induction therapy
- Without Transplant Donor: Patients who did not have transplant donor reported after achieving CR/Cri/leukemia-free state after induction therapy
Arm/Group | With Transplant Donor | Without Transplant Donor
Number analyzed (Participants) | 172 | 214
months | 27.2 [15.3 to NA] — The upper limit of the 95% confidence interval was not calculable because an insufficient number of participants reached the event at the final time point for assessment. | 12.9 [10.3 to 17.0]

4. Secondary Outcome: Disease-free Survival for Maintenance
Description: DFS for maintenance comparison is defined as the time from maintenance randomization until relapse or death of any cause. The censored follow-up time for patients without relapse and death information is the date of last contact. Only patients who remained in CR or CRi after completion of consolidation therapy that were randomized to either observation or decitabine in the maintenance Step were included in this analysis.
Time Frame: Assessed every 3 months for 4 years and then every 6 months for 1 year
Population: Only patients who remained in CR or CRi after completion of consolidation therapy that were randomized to either observation or decitabine in the maintenance step were included in this analysis.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Maintenance : Observation: Patients who remained in CR or CRi after completion of consolidation therapy were randomized to be on observation
- Maintenance : Decitabine: Patients who remained in CR or CRi after completion of consolidation therapy were randomized to receive Decitabine for maintenance therapy.
Arm/Group | Maintenance : Observation | Maintenance : Decitabine
Number analyzed (Participants) | 61 | 59
months | 8.2 [5.1 to 18.7] | 16.3 [10.1 to 26.3]

5. Other Pre Specified Outcome: Expression and Methylation Profiling
Description: DNA methylation profiling and gene expression are evaluated using peripheral blood samples collected at baseline of the maintenance treatment (prior to 2nd randomization). These are to be compared between patients with decitabine and patients on observation.
Time Frame: Baseline of maintenance treatment
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Relapse After Decitabine Maintenance by Epigenetic Signature of Normal Bone Marrow
Description: To examine the epigenetic profiles of remission marrow among patients randomized to observation vs. decitabine to determine whether epigenetic signature of apparently morphologically normal bone marrow is predictive of relapse or response to decitabine maintenance.
  Relapse following complete remission is defined as:
  1. Peripheral Blood Counts
     * Reappearance of blasts in the blood
  2. Bone Marrow Aspirate and Biopsy
     * Presence of > 5% blasts, not attributable to another cause (e.g., bone marrow regeneration).
     * If there are no circulating blasts and the bone marrow contains 5% to 20% blasts, then a repeat bone marrow performed ≥ 1 week later documenting more than 5% blasts is necessary to meet the criteria for relapse.
Time Frame: Assessed every 3 months for 4 years and then every 6 months for 1 year
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Complete Remission Rate by ABC-transporter P-glycoprotein (Pgp)
Description: Patients with all the following are considered as having a complete remission.
  * Peripheral Blood Counts
    1. Neutrophil count > 1.0 x 109 /L
    2. Platelet count ≥ 100 x 109 /L
    3. Reduced hemoglobin concentration or hematocrit has no bearing on remission status
    4. Leukemic blasts must not be present in the peripheral blood
  * Bone Marrow Aspirate and Biopsy
    1. Cellularity of bone marrow biopsy must be > 20% with maturation of all cell lines
    2. < 5% blasts by morphologic review
    3. Auer rods must not be detectable
  * Extramedullary leukemia, such as CNS or soft tissue involvement, must not be present
  The proportion of patients with complete remission will be compared between patients who overexpress Pgp and patients who do not overexpress Pgp.
Time Frame: Assessed every 3 months for 4 years and then every 6 months for 1 year
Reporting Status: Not Posted

8. Other Pre Specified Outcome: To Assess the Intensity of Expression of CXCR4 on Diagnostic Leukemia Cells and to Correlate This Parameter With Other Established Prognostic Factors
Description: Expression of CXCR4 will be assessed in this study by flow cytometric assay. The associations between the expression level and other prognostic factors in patients receiving induction treatment will be evaluated.
Time Frame: Baseline
Reporting Status: Not Posted

9. Other Pre Specified Outcome: The Association Between Somatic Mutations and Relapse
Description: Relapse following complete remission is defined as:
  1. Peripheral Blood Counts
     * Reappearance of blasts in the blood
  2. Bone Marrow Aspirate and Biopsy
     * Presence of > 5% blasts, not attributable to another cause (e.g., bone marrow regeneration).
     * If there are no circulating blasts and the bone marrow contains 5% to 20% blasts, then a repeat bone marrow performed ≥ 1 week later documenting more than 5% blasts is necessary to meet the criteria for relapse.
Time Frame: Assessed every 3 months for 4 years and then every 6 months for 1 year
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Overall Survival by Patient Characteristics and Lifestyle
Description: Overall survival is defined as time from randomization to death or date last known alive. The associations between overall survival and smoking status, obesity, regular acetaminophen use, regular aspirin use, benzene exposure, living in a rural/farm environment and some other underlying exposures and lifestyle factors will be evaluated.
Time Frame: Assessed every 3 months for 4 years and then every 6 months for 1 year
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Copy Number Changes Using Array Comparative Genomic Hybridization (CGH) by Patient Characteristics
Description: Copy number changes will be tested based on array CGH technology. The associations between copy number changes and acute myeloid leukemia patient characteristics will be evaluated.
Time Frame: Baseline
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Quality of Life (QOL) Assessed by Functional Assessment of Cancer Therapy - Leukemia (FACT-Leu)
Description: QOL will be assessed using the Functional Assessment of Cancer Therapy - Leukemia (FACT-Leu). This instrument combines the General version of the Functional Assessment of Cancer Therapy (FACT-G) with a leukemia-specific subscale. The total score of FACT-Leu ranges between 0 and 176. Higher score indicates better QOL.
Time Frame: Assessed at baseline, 14 days after 1st induction treatment, prior to consolidation therapy (day 35-36), prior to maintenance treatment, end of maintenance treatment
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Change in Health-related QOL Over Time
Description: QOL will be assessed using the Functional Assessment of Cancer Therapy - Leukemia (FACT-Leu). This instrument combines the General version of the Functional Assessment of Cancer Therapy (FACT-G) with a leukemia-specific subscale. The total score of FACT-Leu ranges between 0 and 176. Higher score indicates better QOL.
  Changes in QOL will be calculated by subtracting baseline QOL score from follow-up QOL score.
Time Frame: as for outcome 12
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Patient Function Assessed by Functional Assessment of Cancer Therapy - General (FACT-G)
Description: QOL will be assessed using the Functional Assessment of Cancer Therapy - General (FACT-G). FACT-G includes 4 subscales, physical well-being (score range: 0-28), social/family well-being (score range: 0-28), emotional well-being (score range: 0-24), and functional well-being (score range: 0-28). The total score of FACT-G ranges between 0 and 108. Higher score indicates better QOL.
Time Frame: Assessed at baseline
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Change in QOL Post Transplant From Baseline
Description: For those patients who go to allo transplant, the FACT-Leu and the Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-Fatigue) instruments will be administered at the beginning of the conditioning regimen and 100 days (+14 days) post transplant.
  FACT-Leu combines the General version of the Functional Assessment of Cancer Therapy (FACT-G) with a leukemia-specific subscale. The total score of FACT-Leu ranges between 0 and 176. Higher score indicates better QOL.
  FACIT-Fatigue has 13 items and the total score ranges between 0 and 52. Higher score indicates better QOL.
  Changes in QOL will be calculated by subtracting baseline QOL score from follow-up QOL score.
Time Frame: Assessed prior to transplant and 100 days after transplant
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Baseline QOL Scores by Treatment Completion Status
Description: The associations between baseline QOL scores and the ability to finish treatment will be evaluated. Baseline QOL will be assessed using the Functional Assessment of Cancer Therapy - Leukemia (FACT-Leu) and the Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-Fatigue).
  FACT-Leu combines the General version of the Functional Assessment of Cancer Therapy (FACT-G) with a leukemia-specific subscale. The total score of FACT-Leu ranges between 0 and 176. Higher score indicates better QOL.
  FACIT-Fatigue has 13 items and the total score ranges between 0 and 52. Higher score indicates better QOL.
Time Frame: Assessed at baseline
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Assessed every 4 weeks while on treatment and for 30 days after the end of treatment, up to 5 years
Description: All patients enrolled are included in all-cause mortality analysis. Patients who received treatment with adverse event data available are included in AE analysis.
Groups:
- Arm A (Induction: Daunorubicin + Cytarabine): Patients receive daunorubicin intravenously (IV) over 10-15 minutes on days 1-3 and cytarabine IV continuously on days 1-7.
  Patients with residual disease or those who do not achieve an aplastic bone marrow on day 12-14 (i.e., < 5% blasts and < 20% cellularity or markedly/moderately hypocellular) may receive a second course of induction therapy beginning no sooner than day 14.
  Patients who achieve a complete remission (CR) or CR with incomplete marrow recovery (CRi) after induction therapy proceed to consolidation therapy (Cytarabine; Arm C). Patients who achieve a "morphologic leukemia-free state" after induction therapy and who have an HLA-identical donor proceed to consolidation therapy followed by allogeneic stem cell transplantation.
- Arm B (Induction: Clofarabine): Patients receive clofarabine IV over 1 hour on days 1-5. Patients with residual disease or those who do not achieve an aplastic bone marrow on day 12-14 (i.e., < 5% blasts and < 20% cellularity or markedly/moderately hypocellular) may receive a second course of induction therapy beginning no sooner than day 21 and no later than day 56.
  Patients who achieve a complete remission (CR) or CR with incomplete marrow recovery (CRi) after induction therapy proceed to consolidation therapy (Clofarabine; Arm D). Patients who achieve a "morphologic leukemia-free state" after induction therapy and who have an HLA-identical donor proceed to consolidation therapy followed by allogeneic stem cell transplantation.
- Arm C (Consolidation: Cytarabine): Patients in Arm A who achieve a CR or CRi after induction therapy proceed to consolidation therapy (Cytarabine; Arm C). Patients who achieve a "morphologic leukemia-free state" after induction therapy in Arm A and who have an HLA-identical donor proceed to consolidation therapy (Cytarabine; Arm C) followed by allogeneic stem cell transplantation.
  Patients receive cytarabine (consolidation therapy) IV over 1 hour once or twice daily on days 1-6. Treatment repeats every 4-6 weeks for 2 courses.
- Arm D (Consolidation: Clofarabine): Patients in Arm B who achieve a CR or CRi after induction therapy proceed to consolidation therapy (Clofarabine; Arm D). Patients who achieve a "morphologic leukemia-free state" after induction therapy in Arm B and who have an HLA-identical donor proceed to consolidation therapy (Consolidation; Arm D) followed by allogeneic stem cell transplantation.
  Patients receive clofarabine (consolidation therapy) IV over 1 hour on days 1-5. Treatment repeats every 4-6 weeks for 2 courses.
- Arm E (Maintenance: Observation): Patients in Arms C or D who remain in CR or CRi after completion of consolidation therapy are randomized to maintenance therapy (Observation; Arm E).
  Patients undergo observation monthly for 12 months.
- Arm F (Maintenance: Decitabine): Patients in Arms C or D who remain in CR or CRi after completion of consolidation therapy are randomized to maintenance therapy (Decitabine; Arm F).
  Patients receive decitabine IV over 1 hour on days 1-3. Treatment repeats every 4 weeks for 12 months the absence of unacceptable toxicity.
- Arm G (Transplant): Patients in Arms C or D who achieve a CR or CRi or a "morphologic leukemia-free state" after completion of consolidation therapy and who have an HLA-identical donor proceed to allogeneic stem cell transplantation. (Arm G).
  Patients undergo allogeneic peripheral blood stem cell transplantation
Arm/Group | Arm A (Induction: Daunorubicin + Cytarabine) | Arm B (Induction: Clofarabine) | Arm C (Consolidation: Cytarabine) | Arm D (Consolidation: Clofarabine) | Arm E (Maintenance: Observation) | Arm F (Maintenance: Decitabine) | Arm G (Transplant)
All-Cause Mortality (participants affected / at risk) | 284/363 | 295/364 | 0/174 | 0/154 | 0/61 | 0/59 | 0/72
Serious Adverse Events (participants affected / at risk) | 354/356 | 357/360 | 164/170 | 140/148 | 19/59 | 50/54 | 62/70
Other Adverse Events (participants affected / at risk) | 356/356 | 355/360 | 169/170 | 147/148 | 51/59 | 53/54 | 62/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Induction: Daunorubicin + Cytarabine) (N=356) | Arm B (Induction: Clofarabine) (N=360) | Arm C (Consolidation: Cytarabine) (N=170) | Arm D (Consolidation: Clofarabine) (N=148) | Arm E (Maintenance: Observation) (N=59) | Arm F (Maintenance: Decitabine) (N=54) | Arm G (Transplant) (N=70)
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Anemia (Blood and lymphatic system disorders) | 308 | 304 | 118 | 77 | 1 | 9 | 21
Febrile neutropenia (Blood and lymphatic system disorders) | 239 | 199 | 68 | 26 | 0 | 5 | 21
Leukocytosis (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0 | 0 | 1 | 0
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 | 1 | 2 | 0 | 0 | 0 | 0
Blood and lymphatic disorders - Other (Blood and lymphatic system disorders) | 6 | 5 | 1 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 14 | 7 | 2 | 0 | 0 | 0 | 1
Atrial flutter (Cardiac disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Heart failure (Cardiac disorders) | 2 | 4 | 0 | 0 | 0 | 0 | 1
Left ventricular systolic dysfunction (Cardiac disorders) | 7 | 3 | 2 | 2 | 0 | 0 | 0
Mitral valve disease (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Paroxysmal atrial tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pericarditis (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Restrictive cardiomyopathy (Cardiac disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 2 | 5 | 4 | 0 | 0 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 2 | 3 | 0 | 0 | 0 | 0 | 0
Ventricular fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ventricular tachycardia (Cardiac disorders) | 2 | 0 | 1 | 0 | 0 | 0 | 0
Cardiac disorders - Other, specify (Cardiac disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Death NOS (General disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Edema limbs (General disorders) | 3 | 3 | 1 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 25 | 18 | 10 | 4 | 0 | 2 | 3
Fever (General disorders) | 3 | 1 | 4 | 0 | 0 | 0 | 0
Localized edema (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Multi-organ failure (General disorders) | 6 | 4 | 0 | 1 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0
General and administration site - Other (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0
Erythroderma (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Palmar-plantar erythrodysesthesia (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 3 | 0 | 1 | 0 | 0 | 1
Purpura (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 20 | 23 | 3 | 3 | 0 | 0 | 3
Skin ulceration (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Toxic epidermal necrolysis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin and subcutaneous tissue - Other (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Endocrine disorders - Other, specify (Endocrine disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 4 | 0 | 0 | 0 | 0 | 1
Anal hemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 4 | 2 | 0 | 0 | 0 | 1 | 0
Colonic obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 26 | 13 | 7 | 0 | 0 | 2 | 6
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 4 | 1 | 1 | 0 | 0 | 0 | 0
Enterocolitis (Gastrointestinal disorders) | 3 | 3 | 1 | 0 | 0 | 0 | 0
Esophageal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Esophagitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fecal incontinence (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastric hemorrhage (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 0
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Ileal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 2 | 3 | 0 | 1 | 0 | 0 | 0
Mucositis oral (Gastrointestinal disorders) | 13 | 3 | 2 | 1 | 0 | 0 | 5
Nausea (Gastrointestinal disorders) | 8 | 8 | 5 | 0 | 0 | 0 | 5
Oral pain (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0
Rectal fistula (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rectal hemorrhage (Gastrointestinal disorders) | 0 | 2 | 2 | 0 | 0 | 0 | 0
Rectal pain (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Typhlitis (Gastrointestinal disorders) | 8 | 2 | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 4 | 3 | 2 | 0 | 0 | 0 | 2
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Allergic reaction (Immune system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Cytokine release syndrome (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Immune system disorders - Other, specify (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal infection (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Anorectal infection (Infections and infestations) | 0 | 1 | 2 | 0 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bladder infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bone infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bronchial infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Catheter related infection (Infections and infestations) | 15 | 16 | 10 | 3 | 0 | 0 | 0
Encephalitis infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Endocarditis infective (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Endophthalmitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Enterocolitis infectious (Infections and infestations) | 10 | 8 | 3 | 1 | 0 | 0 | 0
Esophageal infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Eye infection (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Gallbladder infection (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Joint infection (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Kidney infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lip infection (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Lung infection (Infections and infestations) | 60 | 42 | 20 | 4 | 0 | 2 | 2
Mucosal infection (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Papulopustular rash (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Peritoneal infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pleural infection (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0 | 1
Rash pustular (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Scrotal infection (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 39 | 27 | 22 | 4 | 0 | 0 | 3
Sinusitis (Infections and infestations) | 2 | 2 | 1 | 0 | 0 | 0 | 0
Skin infection (Infections and infestations) | 8 | 5 | 4 | 2 | 1 | 1 | 1
Small intestine infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Soft tissue infection (Infections and infestations) | 2 | 2 | 2 | 0 | 0 | 0 | 0
Splenic infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Stoma site infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tooth infection (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Upper respiratory infection (Infections and infestations) | 2 | 2 | 0 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 12 | 12 | 1 | 1 | 0 | 2 | 2
Wound infection (Infections and infestations) | 2 | 0 | 2 | 0 | 0 | 0 | 0
Infections and infestations - Other (Infections and infestations) | 25 | 19 | 10 | 4 | 0 | 1 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Prolapse of intestinal stoma (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vascular access complication (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Activated PTT prolonged (Investigations) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 14 | 79 | 7 | 13 | 0 | 1 | 1
Alkaline phosphatase increased (Investigations) | 9 | 6 | 3 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 19 | 80 | 7 | 15 | 0 | 2 | 3
Blood bilirubin increased (Investigations) | 29 | 38 | 7 | 3 | 1 | 0 | 2
CO diffusing capacity decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cardiac troponin I increased (Investigations) | 2 | 0 | 1 | 0 | 0 | 0 | 0
CD4 lymphocytes decreased (Investigations) | 1 | 1 | 0 | 0 | 0 | 0 | 1
Creatinine increased (Investigations) | 12 | 13 | 4 | 1 | 1 | 0 | 3
Ejection fraction decreased (Investigations) | 3 | 0 | 1 | 0 | 0 | 0 | 0
ECG QT corrected interval prolonged (Investigations) | 3 | 1 | 3 | 0 | 0 | 0 | 0
Fibrinogen decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
GGT increased (Investigations) | 1 | 0 | 1 | 2 | 1 | 0 | 0
Hemoglobin increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lipase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 87 | 83 | 44 | 38 | 1 | 4 | 17
Lymphocyte count increased (Investigations) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 343 | 339 | 142 | 124 | 7 | 48 | 45
Platelet count decreased (Investigations) | 346 | 347 | 154 | 126 | 8 | 23 | 40
Urine output decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Weight gain (Investigations) | 2 | 0 | 1 | 0 | 0 | 0 | 0
Weight loss (Investigations) | 5 | 2 | 3 | 1 | 0 | 0 | 0
White blood cell decreased (Investigations) | 349 | 351 | 149 | 126 | 4 | 39 | 52
Investigations - Other, specify (Investigations) | 2 | 4 | 3 | 0 | 0 | 1 | 0
Acidosis (Metabolism and nutrition disorders) | 1 | 2 | 1 | 0 | 0 | 0 | 0
Alkalosis (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 35 | 15 | 6 | 1 | 0 | 0 | 7
Dehydration (Metabolism and nutrition disorders) | 8 | 2 | 5 | 4 | 0 | 0 | 1
Glucose intolerance (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 2
Hyperglycemia (Metabolism and nutrition disorders) | 17 | 11 | 11 | 0 | 0 | 2 | 6
Hyperkalemia (Metabolism and nutrition disorders) | 2 | 1 | 1 | 0 | 0 | 0 | 1
Hypermagnesemia (Metabolism and nutrition disorders) | 7 | 4 | 0 | 0 | 0 | 0 | 1
Hypernatremia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hyperuricemia (Metabolism and nutrition disorders) | 3 | 0 | 1 | 1 | 0 | 0 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 9 | 9 | 4 | 0 | 0 | 0 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 21 | 19 | 1 | 0 | 0 | 0 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypokalemia (Metabolism and nutrition disorders) | 24 | 28 | 3 | 6 | 0 | 1 | 2
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 3
Hyponatremia (Metabolism and nutrition disorders) | 23 | 14 | 5 | 2 | 0 | 1 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 37 | 26 | 1 | 2 | 0 | 0 | 1
Tumor lysis syndrome (Metabolism and nutrition disorders) | 5 | 3 | 0 | 0 | 0 | 0 | 0
Metabolism and nutrition - Other (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 2 | 0 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 1 | 0 | 0 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 14 | 9 | 8 | 0 | 0 | 1 | 1
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2 | 0 | 0 | 0 | 0
Musculoskeletal and connective - Other (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ataxia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cognitive disturbance (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 2 | 0 | 0 | 0
Encephalopathy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 3 | 3 | 1 | 0 | 0 | 0 | 1
Intracranial hemorrhage (Nervous system disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Leukoencephalopathy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Stroke (Nervous system disorders) | 1 | 3 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 5 | 4 | 2 | 0 | 0 | 0 | 0
Vasovagal reaction (Nervous system disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Neoplasms - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Conjunctivitis (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Eye pain (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Eyelid function disorder (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Uveitis (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vitreous hemorrhage (Eye disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Eye disorders - Other, specify (Eye disorders) | 1 | 0 | 1 | 0 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Confusion (Psychiatric disorders) | 5 | 3 | 2 | 0 | 0 | 0 | 1
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 6 | 2 | 0 | 0 | 0 | 0 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0 | 0 | 0 | 0 | 0
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 23 | 20 | 4 | 2 | 0 | 1 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 | 8 | 1 | 0 | 0 | 0 | 2
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 18 | 18 | 2 | 0 | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 8 | 5 | 1 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 14 | 9 | 1 | 0 | 0 | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory thoracic mediastinal - Other (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 14 | 15 | 3 | 0 | 0 | 0 | 1
Chronic kidney disease (Renal and urinary disorders) | 2 | 1 | 2 | 0 | 0 | 0 | 0
Hematuria (Renal and urinary disorders) | 3 | 1 | 0 | 0 | 0 | 0 | 0
Renal and urinary disorders - Other (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Scrotal pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Testicular disorder (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Capillary leak syndrome (Vascular disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0
Hematoma (Vascular disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 15 | 12 | 7 | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 19 | 18 | 8 | 2 | 0 | 0 | 1
Thromboembolic event (Vascular disorders) | 5 | 3 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Induction: Daunorubicin + Cytarabine) (N=356) | Arm B (Induction: Clofarabine) (N=360) | Arm C (Consolidation: Cytarabine) (N=170) | Arm D (Consolidation: Clofarabine) (N=148) | Arm E (Maintenance: Observation) (N=59) | Arm F (Maintenance: Decitabine) (N=54) | Arm G (Transplant) (N=70)
Anemia (Blood and lymphatic system disorders) | 327 | 327 | 162 | 141 | 40 | 48 | 59
Alanine aminotransferase increased (Investigations) | 161 | 255 | 77 | 79 | 6 | 12 | 24
Alkaline phosphatase increased (Investigations) | 151 | 166 | 78 | 60 | 9 | 7 | 16
Aspartate aminotransferase increased (Investigations) | 179 | 262 | 72 | 75 | 5 | 14 | 22
Blood bilirubin increased (Investigations) | 159 | 213 | 57 | 44 | 3 | 9 | 13
Creatinine increased (Investigations) | 102 | 93 | 29 | 24 | 4 | 10 | 16
Neutrophil count decreased (Investigations) | 193 | 196 | 93 | 85 | 11 | 45 | 36
Platelet count decreased (Investigations) | 285 | 283 | 156 | 134 | 36 | 50 | 51
White blood cell decreased (Investigations) | 252 | 267 | 143 | 121 | 29 | 51 | 46
Hypermagnesemia (Metabolism and nutrition disorders) | 49 | 42 | 7 | 10 | 0 | 0 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 140 | 122 | 77 | 47 | 6 | 6 | 36

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-27): https://cdn.clinicaltrials.gov/large-docs/08/NCT02085408/Prot_SAP_000.pdf